CLINICAL TRIAL: NCT06436417
Title: Monitoring Functional Capacity Through Heart Rate Variability Within the Multimodal Rehabilitation Program in Adult Surgery
Brief Title: Functional Capacity Through HRV in Multimodal Rehabilitation for Adult Surgery
Acronym: PreANI
Status: Recruiting | Type: Observational
Sponsor: Investigation Group Anesthesia, Resuscitation, And Perioperative Medicine of Aragon (Network)
Responsible Party: Sponsor
Other Study IDs: PreANI001
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Frailty in Adult Surgery
Keywords: Heart rate variability, prehabilitation, major surgery, frailty, physiological reserve
MeSH Terms: conditions — Frailty | interventions — Monitoring, Physiologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Patients who do not undergo prehabilitation.
  Interventions: Device: Analgesia Nociception Index (ANI) Monitor
- Prehabilitation: Patients who undergo trimodal prehabilitation including physical exercise, nutritional supplementation, and psychological support.
  Interventions: Device: Analgesia Nociception Index (ANI) Monitor; Behavioral: Trimodal Prehabilitation

INTERVENTIONS:
Device: Analgesia Nociception Index (ANI) Monitor — Non-invasive monitoring of HRV to evaluate autonomic nervous system activity using the indices of Energy (SDNN) and ANI (HFnu).
Behavioral: Trimodal Prehabilitation — Program of physical exercise, nutritional supplementation, and psychological support according to the RICA guidelines of the Spanish Group for Multimodal Rehabilitation.
  Groups: Prehabilitation

SUMMARY:
This prospective, observational cohort study investigates heart rate variability (HRV) monitoring using the Analgesia Nociception Index (ANI) monitor in adult patients undergoing major surgery within a multimodal rehabilitation program. The objective is to correlate HRV indices with functional capacity, physiological reserve, and frailty during the prehabilitation phase.

DETAILED DESCRIPTION:
The study evaluates HRV using the ANI monitor to determine adaptation to training load, optimize analgesic and anesthetic dosing, and predict postoperative complications. The HRV indices of Energy (SDNN) and ANI (HFnu) are monitored at two points: the initial pre-anesthesia consultation and one week before surgery. Results will be compared with the 6-minute walk test, MUST nutrition screening scale, and clinical frailty and FRAIL scales.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Scheduled for major adult surgery
* Any ASA classification
* Signed informed consent

Exclusion Criteria:

* Urgent surgery
* Severe cognitive impairment
* Patient refusal to participate
* Pediatric patients
* Cardiac arrhythmia or atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing major surgery within a multimodal rehabilitation program in various hospitals in Spain.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of HRV indices with functional capacity and frailty | From initial pre-anesthesia consultation to 30 days postoperatively
  Evaluation of the correlation between HRV indices (Energy and ANI) and current parameters used to assess functional capacity, physiological reserve, and frailty.

SECONDARY OUTCOMES:
Reduction of postoperative complications | 30 days postoperatively
  Evaluation of the relationship between higher preoperative functional reserve and lower number of complications, mortality, and hospital stay at 30 days postoperatively.
Intraoperative decisions based on HRV | During the perioperative period
  Analysis of whether HRV monitoring guides the workload during prehabilitation and the titration of drugs during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Aragón-Benedí, M.D., Ph.D.,, Study Chair — Miguel Servet University Hospital
Locations (1):
- Miguel Servet University Hospital, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data (IPD) with other researchers.